CLINICAL TRIAL: NCT06800417
Title: Performance and Safety of the Innofix® Screw as Part of Stabilization of a Non-displaced Pathologic Fracture (Complete or Impending) of the Pelvic Bone of Cancer Patients by Mini-invasive Percutaneous Fixation by Internal Cemented Screw
Brief Title: Performance and Safety of the Innofix® Screw (IF25)
Acronym: IF25
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Innoprod Medical (Industry)
Collaborators: EVAMED (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IF25; 2025-A00016-43 (Registry Identifier: French clinical trials database [ANSM])
Record Dates: First submitted 2025-01-17; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Pathologic Fracture
Keywords: FICS; Pelvis; Cancer
MeSH Terms: conditions — Fractures, Spontaneous; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult cancer patient with a non-displaced pelvic pathologic fracture (Experimental): The fracture of the patients, treated with InnoFix® screw, is stabilized with a percutaneous fixation by internal cemented screw. This procedure is carried out by mini-invasive approach.
  Interventions: Device: Percutaneous fixation by internal cemented screw (InnoFix®)

INTERVENTIONS:
Device: Percutaneous fixation by internal cemented screw (InnoFix®) — Percutaneous fixation by internal cemented screw

SUMMARY:
The purpose of this clinical investigation is to collect data about the safety and the performances of the InnoFix® screw : Clinical performances (Pain reduction due to the fracture treatment, maintenance of the stabilizaton of the treated fracture and mobility improvement) / Technical performances (Percutaneous implantation by mini-invasive approach, Efficiency of percutaneous implementation and efficiency of percuatneous cementing) / Safety performances (Preservation of the screw stability after implantation and preservation of the screw integrity after implantation). The safety and performance data about the InnoFix® screw will be used to obtain their CE marking according to the regulation (EU) 2017/745.

The principal objective of this clinical investigation is to assess the postoperative reduction in pain level of the patient at 6 weeks follow-up.

ELIGIBILITY:
Inclusion Criteria:

* The patient is 18 years old or more
* The patient is a cancer patient
* The patient needs a stabilization of a non-displaced pathologic fracture (complete or impending) of the pelvic bone
* The patient is symptomatic with musculoskeletal pain exacerbated during movement or weight bearing
* The patient has been informed and he has signed the informed consent
* The patient must be willing and able to comply with all study requirements including follow-up visits and radiographic assessments
* The patient is affiliated with the French social security system

Exclusion Criteria:

* The patient has got a displaced fracture or an unstable fracture justifying conventional surgical fixation
* The patient is a pregnant woman or considered getting pregnant during its investigation participation
* The patient presents medical conditions that could have an impact on the clinical investigation (under responsibility of the investigator)
* The patient has got one or more contraindications to general anaesthesia
* The patient has got an insufficient bone strength (severe osteoporosis, local infection, or tumor osteolysis) precluding a correct and long-term fixation
* The use of the InnoFix® screw can interfere with anatomical structures or physiological performances
* The patient has got an insufficient tissue coverage at the surgical site
* The patient has got a sepsis, fever, subcutaneous or cutaneous infection on the implantation way, deep abscess in contact with the fracture site
* The patient has got a mental or neuromuscular disorder that may cause fixation failure or postoperative complications
* The patient is allergic and/or hypersensitive to a component of the InnoFix® modules, of the InnoTool™ instruments and to the used cement
* The patient has got a haemostasis disorder ((INR >1.5, platelets <50x109/L)
* The patient participates to another clinical investigation
* The patient's life expectancy is lower than 6 months
* The patient is under guardianship, curatorship or legal protection
* The patient is deprived of liberty by a judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Rate of patients which have a pain reduction rate, at 6 weeks postoperatively, equal or superior to 30% | From the patient inclusion date to 6 weeks postoperatively
  Pain reduction is measured with the VAS scale : Zero is equivalent to no pain and 10 indicates the worst possible pain

SECONDARY OUTCOMES:
Rate of patients which have a pain reduction rate, at 6 months postoperatively, equal or superior to 30% | From the patient inclusion date to 6 months postoperatively
  The pain is measured with the VAS scale: Zero is equivalent to no pain and 10 indicates the worst possible pain
Rate of postoperative stable fractures | From end surgery to 6 weeks and 6 months postoperatively
  Fracture stability is assessed with medical imaging: Length of fracture line in millieter (complete fracture) or fracture occurernce (impending fracture)
Rate of patients which have a mobility improvement rate postoperatively | From the patient inclusion date to 6 weeks and 6 months postoperatively
  Mobility is measured with ECOG scale:
Implantation success rate of the InnoFix® screw | At the end of surgery
  Implantation succes is measured with medical imaging: Screw position compared to the fracture line and distance, in millimeters, of the distal tip of screw compared to the planned area and protrusion, in millimeters, of the proximal part of screw from the external cortex
Satisfaction rate of the radiologist regarding the efficiency of the percutaneous implementation | At the end of surgery
  Efficiency of percutaneous implementation is based on the experiency of the radaiologist
Satisfaction rate of the radiologist regarding the efficiency of the percutaneous cementing | At the end of surgery
  Efficiency of percutaneous cementing is based on the experiency of the radaiologist
Rate of stable InnoFix® screws postoperatively | From end surgery to 6 weeks and 6 months postoperatively
  Screw stability is measured with medical imaging: Screw displacement in millimeters and contact with anatomical structures or other implanted devices
Rate of InnoFix® screws with their integrity preserved postoperatively | From end surgery to 6 weeks and 6 months postoperatively
  Screw integrity is measured with medical imaging: Disassembly, breakage or bending in millimeters
Rate of patient which have had, at least, one adverse event in relation with the InnoFix® screw postoperatively | From the patient inclusion date to 6 months postoperatively
  Adverse event reported
Rate of patient which have had, at least, one serious adverse event in relation with the InnoFix® screw postoperatively | From the patient inclusion date to 6 months postoperatively
  Serious adverse event reported

CONTACTS AND LOCATIONS:
Overall Officials: Lambros TSELIKAS, Principal Investigator — Gustave ROUSSY Cancer Institute - Villejuif; Xavier BUY, Principal Investigator — BERGONIE Institute - Bordeaux; Roberto Luigi CAZZATO, Principal Investigator — Strasbourg Civil Hospital - Strasbourg

IPD SHARING:
Plan to Share IPD: No
Sponsor commitment to not transfert data outside the European Union